CLINICAL TRIAL: NCT05581433
Title: Vapocoolant Spray Application During Intraarticular Knee Injection: Myth or Reality? A Prospective Randomized Controlled Trial
Brief Title: Vapocoolant Spray Application During Intraarticular Knee Injection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istanbul Rumeli University (Other)
Responsible Party: Principal Investigator, Cagdas PAMUK, Asisstant Professor, Istanbul Rumeli University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: E-10840098-772.02-762
Record Dates: First submitted 2022-10-11; First posted 2022-10-14 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2022-10

CONDITIONS: Osteo Arthritis Knee; Injection Site Discomfort; Injection Fear
MeSH Terms: conditions — Iatrophobia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- vapocoolan spray applied group before injection (Active Comparator): Vapocoolant spray will be applied to patients in this group before intra-articular knee injection.
  Interventions: Other: Topical Cooling Spray
- placebospray applied group before injection (Placebo Comparator): Placebo spray will be applied to patients in this group before intra-articular knee injection.
  Interventions: Other: Saline spray as Placebo
- No administration group before injection (No Intervention): In this group, no pain reliever application will be made before the application.

INTERVENTIONS:
Other: Topical Cooling Spray — The process of cooling the area to be injected with a cooling spray before the application in order to reduce the pain.
  Arms: vapocoolan spray applied group before injection
Other: Saline spray as Placebo — Application of saline spray without cooling effect to the area to be injected for placebo purposes
  Arms: placebospray applied group before injection

SUMMARY:
The goal of this observational study is to learn about the effects of vapocoolant spray applied during intraarticular knee injections on pain and anxiety compared to injections without any agent application in patients with knee osteoarthritis.

The main questions it aims to answer are: • Contrary to popular belief, does coolant spray application really reduce pain? • Does it have an advantage over patients with placebo or no spray at all? After intraarticular knee hyaluronic acid application, patients will be asked to indicate injection-related pain and anxiety levels on a 100mm visual analog scale. Researchers will compare the patient groups who were applied coolant spray, placebo spray and injection without any spray.

DETAILED DESCRIPTION:
Patients who underwent intra-knee hyaluronic acid injection due to knee degenerative diseases (osteoarthritis), meniscus and cartilage problems between October 2022 and December 2022 will be prospectively included in the study. Demographic characteristics of the patients (age, gender, body mass index), degree of knee degeneration, and past surgical procedures will be recorded.

Before intra-articular injection can be given, one group will be sprayed with a vapocoolant, and one group will receive a placebo spray, while another group will receive no analgesic treatment while injection. Which patient will be evaluated in which group will be decided by randomization on the website www.random.org.

1 minute after the injection, the patients will be asked to indicate their pain level (1) and anxiety level (2) while inserting the needle on the 100mm Visual Analogue Scale (VAS). The same survey will be repeated after 10 minutes, and whether they are satisfied with the whole process will be measured with the same scale and the results will be recorded. The results will be compared between the groups, and the demographic characteristics of the patients, the level and types of disease, and the effects of vapocoolant spray application will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* The patients with osteoarthritis of the knee undergoing a normal HA injection scheduled between October 2022 and December 2022.

Exclusion Criteria:

* Prior history of injection of the knee joint
* Inability to understand the Visual Analog Scale,
* History of cold intolerance
* Use of pain medications or topical anesthetics within the previous 24 hours
* Abnormal sensation or signs of infection over the injection site.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-10-20 (Actual); Primary Completion 2022-10-20 (Actual); Study Completion 2023-01-30 (Estimated)

PRIMARY OUTCOMES:
pain during injection | 10 seconds
  the level of pain felt when the needle is inserted

SECONDARY OUTCOMES:
patient satisfaction level | 10 minutes
  patient satisfaction level due to the application

CONTACTS AND LOCATIONS:
Overall Officials: Çağdaş Pamuk, MD, Principal Investigator — Istanbul Rumeli University
Locations (1):
- Private Silivri Anadolu Hospital, Istanbul, Silivri, Turkey (Türkiye)